CLINICAL TRIAL: NCT00560027
Title: Screening, Referral and Case Management for Postpartum Depression and Intimate Partner Violence in an Urban Pediatric Practice
Brief Title: Case Management Study for Postpartum Depression and Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Leonard & Helen R. Stulman Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Barry Solomon, Associate Professor of Pediatrics, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20064046
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Postpartum Depression; Intimate Partner Violence
Keywords: postpartum depression; intimate partner violence
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Case Management by Family Support Counselor (not RCT) — N/A. Had planned to study RCT of case management intervention but unable to carry out RCT. Instead studied screening practice and healthcare utilization in mothers with PPD, IPV or both.

SUMMARY:
The objective of the study was to assess the prevalence, timing, and co-occurrence of positive screens for maternal postpartum depression (PPD) and intimate partner violence (IPV) for women bringing their young infants for pediatric primary care and examine relationships between PPD, IPV and children's healthcare utilization from birth to 2 years.

DETAILED DESCRIPTION:
Post-partum depression (PPD) and intimate partner violence (IPV) negatively affect the health and well-being of millions of women each year. In turn, PPD and IPV frequently compromise women's ability to form a strong mother-infant bond, which potentially impacts their children's health and well-being. Limited information exists regarding the prevalence of PPD, IPV, and the co-occurrence of the two. Similarly, empirically tested interventions designed to improve outcomes for these women and their infants are lacking.

The objective of the research was to assess the prevalence, timing, and co-occurrence of positive screens for maternal postpartum depression and intimate partner violence and examine their relationships with children's healthcare utilization from birth to 2 years.

As per routine protocol in the Harriet Lane Clinic (HLC), all mothers bringing their infants for a well baby visit (birth to 6 month visit) are screened for PPD and IPV using a brief, self-administered paper-based questionnaire at the start of the visit. Appropriate resource and referral materials will be provided by a Family Support Counselor (FSC) in the clinic. Between February and March 2008, mothers bringing newborn, 2-, 4-, or 6-month-old children to an urban primary care clinic were screened for postpartum depression and intimate partner violence. A retrospective chart review abstracted demographic data, maternal responses on the postpartum depression/intimate partner violence screen at the initial and subsequent visits, and, from the child's birth to second birthday, adherence with well-child care and use of pediatric acute care and emergency department visits. Descriptive, bivariate, and multivariate analyses were conducted.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking mothers of infants presenting for their newborn, two, four or six month visits to their primary care provider in the Harriet Lane Clinic

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Positive screens for PPD and/or IPV | 12 months

SECONDARY OUTCOMES:
Healthcare utilization over 2 years (acute care, emergency and well visits) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Solomon, MD, MPH, Principal Investigator — Johns Hopkins University; Megan Bair-Merritt, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Harriet Lane Clinic, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kornfeld BD, Bair-Merritt MH, Frosch E, Solomon BS. Postpartum depression and intimate partner violence in urban mothers: co-occurrence and child healthcare utilization. J Pediatr. 2012 Aug;161(2):348-53.e2. doi: 10.1016/j.jpeds.2012.01.047. Epub 2012 Mar 8. PMID 22404952